CLINICAL TRIAL: NCT04185987
Title: Evaluation of the Contamination of Elastomeric Ligatures
Brief Title: Evaluation of the Contamination of Ligatures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Aysegul Gulec, Principal investigator, University of Gaziantep
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017/169
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Orthodontics
Keywords: bacterial adhesion; elastomeric ligatures

STUDY DESIGN:
Intervention Model Description: 2 a cross-over, in vivo study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microbial colonisation (Experimental): microbial sample collection was done at the end of the time periods T1 (6 weeks after bonding ), 10 weeks after bonding (T2), 14 weeks after bonding (T3), 18 weeks after bonding (T4)
  Interventions: Other: Leone slide low friction elastomeric ligature; Other: RMO tough - o energy elastomeric ligature; Other: Dentsply sili tie elastomeric ligature; Other: AO twisted ended ligature wire
- Plaque index (Experimental): Plaque index was measured prior to bonding (T0), 6 weeks after bonding (T1),10 weeks after bonding (T2), 14 weeks after bonding (T3), 18 weeks after bonding (T4)
  Interventions: Other: Leone slide low friction elastomeric ligature; Other: RMO tough - o energy elastomeric ligature; Other: Dentsply sili tie elastomeric ligature; Other: AO twisted ended ligature wire
- Gingival index (Experimental): Gingival index was measured prior to bonding (T0), 6 weeks after bonding (T1), 10 weeks after bonding (T2), 14 weeks after bonding (T3), 18 weeks after bonding (T4)
  Interventions: Other: Leone slide low friction elastomeric ligature; Other: RMO tough - o energy elastomeric ligature; Other: Dentsply sili tie elastomeric ligature; Other: AO twisted ended ligature wire
- surface roughness (Experimental): surface roughness was measured before usage and after 4-weeks usage
  Interventions: Other: Leone slide low friction elastomeric ligature; Other: RMO tough - o energy elastomeric ligature; Other: Dentsply sili tie elastomeric ligature; Other: AO twisted ended ligature wire

INTERVENTIONS:
Other: Leone slide low friction elastomeric ligature — Leone slide low friction elastomeric ligature application
Other: RMO tough - o energy elastomeric ligature — RMO tough - o energy elastomeric ligature application
Other: Dentsply sili tie elastomeric ligature — Dentsply sili tie elastomeric ligature application
Other: AO twisted ended ligature wire — AO twisted ended ligature wire application

SUMMARY:
This crossover, in-vivo study was carried out with 10 patients who have been started to be treated at Orthodontics Department. 3 elastomeric ligatures were examined in terms of microbiological and surface roughness.

DETAILED DESCRIPTION:
The development of dental plaque has been associated with several environmental and individual factors including diet composition, oral hygiene, the quality of saliva, the composition of the oral microflora and immune factors. Orthodontic fixed appliances also impede the maintenance of oral hygiene. Plaque accumulation surrounding orthodontic appliances leads to enamel demineralization caused by organic acids produced by bacteria in the dental plaque.

In patients with fixed orthodontic treatment, common pathological changes are gingivitis, bleeding and gingival growth; thus, gingival index and plaque index parameters have been used as indicators of periodontal disease in many studies. Enamel demineralization which results in white spot formation is observed due to the increase in the number and volume of acid-producing bacteria, and the decrease in pH level because of the glucose metabolized by these cariogenic bacteria . The most commonly investigated bacteria among those mentioned above is Streptococcus Mutans. In the literature, it has been the subject of many studies, including those investigating the correlation between the S. mutans count and the amount of adhesive left between brackets and the enamel, adhesion of S. mutans to nickel titanium and copper-nickel brackets, the difference in S. mutans colonization between self-ligation system and normal brackets, and the effect of elastomeric rings and ligature wires on S. mutans colonization.

Non-conventional elastomeric ligatures were produced in order to reduce the friction of orthodontic sliding mechanics. Manufacturers claim that non-conventional elastomeric ligatures reduced ligation friction by 60% compared to conventional modules. It was reported in another study that brackets combined via non-conventional elastomeric ligatures resulted in a reduced friction force compared to conventional elastomeric ligatures in any wires from 14-inch NITI to 19.25 SS.

To our current knowledge, bacterial colonization on non-conventional elastomeric ligatures was investigated in one study only, using microbial culture technique. In light of this information, present study was aimed to compare S. mutans colonization among different commercial types of non-conventional ligatures and ligature wires. The surface structures of these ligature types also will be investigated by atomic force microscope (AFM) and the results of this investigation will be associated with the results of bacterial colonization amount.

ELIGIBILITY:
Inclusion Criteria:

* permanent teeth in the mouth
* patients with good oral hygiene
* patients did not use antimicrobial drugs such as antibiotics and mouthwashes 3 weeks before the study period and within the 18-week period covering the study period.

Exclusion Criteria:

* smoker

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Microbial colonisation change of S mutans | up to 18 weeks
  Measurement of microbial colonisation change of the interventions with real time PCR
surface roughness identification with atomic force microscope | up to 4 weeks
  measurement of surface roughness identification of the interventions by atomic force microscope

SECONDARY OUTCOMES:
Plaque index | through study completion, 18 weeks
  Measurement of plaque index

OTHER OUTCOMES:
Gingival index | through study completion, 18 weeks
  Measurement of gingival index

CONTACTS AND LOCATIONS:
Overall Officials: Çağlar Dağdeviren, Study Chair — University of Gaziantep; Fahriye Ekşi, Study Chair — University of Gaziantep; Mustafa sağlam, Study Chair — University of Gaziantep; Mehmet Kahraman, Study Chair — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)